CLINICAL TRIAL: NCT04162522
Title: Integrated Biological Markers for the Prediction of Treatment Response in Depression: Validation Study
Brief Title: Canadian Biomarker Integration Network for Depression (CAN-BIND) - Validation Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Unity Health Toronto (Other); Baycrest (Other); Centre for Addiction and Mental Health (Other); McMaster University (Other); Queen's University (Other); University of Ottawa (Other); University of British Columbia (Other); University of Calgary (Other); McGill University (Other); Dalhousie University (Other); University of Michigan (Other); Simon Fraser University (Other)
Responsible Party: Principal Investigator, Sidney Kennedy, Professor of Psychiatry, University of Toronto, Arthur Sommer Rotenberg Chair in Suicide & Depression Studies, St. Michael's Hospital, Principal Investigator, Canadian Biomarker Integration Network for Depression, University Health Network, University Health Network, Toronto
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-5371
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Major Depressive Disorder
Keywords: major depression; major depressive disorder; MDD; escitalopram; brexpiprazole; neuroimaging; genomics; proteomics; metabolomics
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram; Dexetimide; brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- escitalopram (10-20 mg) (Active Comparator): Participants are given escitalopram for 8 weeks. At week 8, participants will be assessed and classified as "responders" or "non-responders". Responders will continue on escitalopram until the study endpoint (16 weeks).
  Interventions: Drug: Escitalopram
- brexpiprazole (0.5-2 mg) (Active Comparator): At week 8, participants classified as "non-responders" will be given 8 weeks of brexpiprazole as add-on treatment to escitalopram.
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Escitalopram — Participants are given escitalopram for 8 weeks. At week 8, those classified as responders will continue on escitalopram until the end of study.
  Other Names: Cipralex
  Arms: escitalopram (10-20 mg)
Drug: Brexpiprazole — Participants who are classified as non-responders are given 8 weeks add-on brexpiprazole, in addition to escitalopram, for the remainder of the study.
  Other Names: Rexulti
  Arms: brexpiprazole (0.5-2 mg)

SUMMARY:
This is a validation study that will replicate a completed study designed to assess biomarkers of treatment response to standard antidepressant treatment. The goal of this study is to integrate clinical, imaging, EEG, and molecular data across 8 sites to predict treatment outcome for patients experiencing a major depressive episode (MDE).

DETAILED DESCRIPTION:
This is a multi-site study to replicate a previous multi-site, multi-platform study completed by the Canadian Biomarker Integration Network in Depression (CAN-BIND). This study aims to validate the integrated array of markers of response and non-response to first line antidepressant treatments that were previously identified in the original aforementioned study. This will be accomplished through collection of clinical, neurophysiological, and molecular measures. This is not a study to evaluate efficacy of medications; medications in this study have been approved by Health Canada and are widely used for the treatment of MDD.

In this study, individuals diagnosed with MDD in a current major depressive episode (MDE) will be treated with open-label escitalopram for 8 weeks. At week 8, participants will be assessed for treatment response (defined as a ≥50% reduction in Montgomery Asberg Depression Rating Scale score). Responders will continue on escitalopram for 8 more weeks. Non-responders will be given add-on brexpiprazole treatment, in addition to escitalopram, for 8 weeks.

Over the 16 weeks, pariticipants will attend 7 clinical visits where they will complete clinical assessments (clinician administered and self-report) and cognitive tests; provide blood, urine, and stool samples; undergo neuroimaging procedures (MRI and EEG); and provide speech samples. At the end of the study, modeling methods will be used to integrate data from these measures to determine the features that best predict treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients 18 to 60 years of age.
* Meet DSM-5 criteria for MDE in MDD as determined by the MINI.
* Episode duration > 3 months.
* Free of psychotropic medications for at least 5 half-lives (e.g. 1 week for most antidepressants, 5 weeks for fluoxetine) before baseline Visit 1.
* MADRS score ≥ 24.
* Fluency in English, sufficient to complete the interviews and self-report questionnaires.

Exclusion Criteria:

* Any diagnosis, other than MDD, that is considered the primary diagnosis.
* Bipolar I or Bipolar-II diagnosis.
* Presence of a significant Axis II diagnosis (borderline, antisocial).
* High suicidal risk, defined by clinician judgment.
* Substance dependence/abuse in the past 6 months.
* Presence of significant neurological disorders, head trauma, or other unstable medical conditions.
* Pregnant or breastfeeding.
* Failure of 4 or more adequate pharmacologic interventions (as determined by the Antidepressant Treatment History Form).
* Started psychological treatment within the past 3 months with the intent of continuing treatment.
* Patients who have previously failed escitalopram or showed intolerance to escitalopram or brexpiprazole, and patients at risk for hypomanic switch (i.e. with a history of antidepressant induced hypomania).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Montgomery Asberg Depression Rating Scale (MADRS) scores from baseline | Week 8, Week 16
  Measured as clinical response, defined as a decrease in Montgomery Asberg Depression Rating Scale (MADRS) score at the Week 8 and Week 16 visits, by 50% or greater, from MADRS score at Baseline visit (i.e., lower MADRS scores = better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Sidney H Kennedy, MD, Principal Investigator — University Health Network, St. Michael's University, University of Toronto
Locations (6):
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - McMaster University, Hamilton, Ontario
  - Queen's University, Kingston, Ontario
  - University Health Network, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
This study is funded by the Ontario Brain Institute (OBI). Data collected from this study is entered into a research database called "Brain-CODE", deployed at a High Performance Computer Virtual Lab (HPCVL). The HPCVL supports the regulatory-compliant (e.g. 21 CRF Part 11, HIPPA, PIPEDA) processes for securing privacy of healthcare data.

REFERENCES:
- [Background] Lam RW, Milev R, Rotzinger S, Andreazza AC, Blier P, Brenner C, Daskalakis ZJ, Dharsee M, Downar J, Evans KR, Farzan F, Foster JA, Frey BN, Geraci J, Giacobbe P, Feilotter HE, Hall GB, Harkness KL, Hassel S, Ismail Z, Leri F, Liotti M, MacQueen GM, McAndrews MP, Minuzzi L, Muller DJ, Parikh SV, Placenza FM, Quilty LC, Ravindran AV, Salomons TV, Soares CN, Strother SC, Turecki G, Vaccarino AL, Vila-Rodriguez F, Kennedy SH; CAN-BIND Investigator Team. Discovering biomarkers for antidepressant response: protocol from the Canadian biomarker integration network in depression (CAN-BIND) and clinical characteristics of the first patient cohort. BMC Psychiatry. 2016 Apr 16;16:105. doi: 10.1186/s12888-016-0785-x. PMID 27084692
- [Background] Kennedy SH, Lam RW, Rotzinger S, Milev RV, Blier P, Downar J, Evans KR, Farzan F, Foster JA, Frey BN, Giacobbe P, Hall GB, Harkness KL, Hassel S, Ismail Z, Leri F, McInerney S, MacQueen GM, Minuzzi L, Muller DJ, Parikh SV, Placenza FM, Quilty LC, Ravindran AV, Sassi RB, Soares CN, Strother SC, Turecki G, Vaccarino AL, Vila-Rodriguez F, Yu J, Uher R; CAN-BIND Investigator Team. Symptomatic and Functional Outcomes and Early Prediction of Response to Escitalopram Monotherapy and Sequential Adjunctive Aripiprazole Therapy in Patients With Major Depressive Disorder: A CAN-BIND-1 Report. J Clin Psychiatry. 2019 Feb 5;80(2):18m12202. doi: 10.4088/JCP.18m12202. PMID 30840787
- [Background] Kennedy SH, Downar J, Evans KR, Feilotter H, Lam RW, MacQueen GM, Milev R, Parikh SV, Rotzinger S, Soares C. The Canadian Biomarker Integration Network in Depression (CAN-BIND): advances in response prediction. Curr Pharm Des. 2012;18(36):5976-89. doi: 10.2174/138161212803523635. PMID 22681173
- See also: CAN-BIND study website — http://www.canbind.ca
- See also: Maclean's news article on suicide prediction and CAN-BIND research — http://www.macleans.ca/society/how-ai-is-helping-to-predict-and-prevent-suicides/